CLINICAL TRIAL: NCT01646762
Title: Phase II Trial of Nab-paclitaxel (Abraxane®) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not pass the Stage 1 interim analysis.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1182; NCI-2012-00879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-007291; MC1182 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2012-07-20 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2016-12

CONDITIONS: Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with multiple myeloma that has returned or did not respond to treatment. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy (overall response rate) of single agent nab-paclitaxel (Abraxane) (paclitaxel albumin-stabilized nanoparticle formulation) in patients with relapsed or refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the adverse events associated with use of single agent nab-paclitaxel (Abraxane) in patients with relapsed or refractory multiple myeloma.

II. To evaluate overall survival, time to progression, and duration of response among patients with relapsed or refractory multiple myeloma undergoing treatment with single agent nab-paclitaxel (Abraxane).

OUTLINE:

Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count >= 500/mm^3
* Platelet count >= 25000/mm^3
* Hemoglobin >= 6 g/dL
* Total bilirubin =< 2.5 X institutional upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 5 X ULN
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5 X ULN
* Creatinine =< 3 mg/dL
* Patients with relapsed or refractory myeloma who have had >= 3 lines of prior therapy
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Ability to understand and the willingness to sign a written informed consent document
* Negative (serum) pregnancy test done =< 7 days prior to registration, for women of childbearing potential only; NOTE: Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Willing to return to enrolling institution (Mayo Clinic in Arizona) for follow-up and all study treatments

Exclusion Criteria:

* Myelosuppressive therapy for myeloma =< 14 days prior to registration or those who have not recovered from acute reversible adverse events due to agents administered > 21 days earlier
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are allowed while on protocol treatment; patients may be receiving stable doses of corticosteroids with a maximum dose of 10 mg of prednisone per day if they are being given for disorders other than lymphoma such as rheumatoid arthritis, polymyalgia rheumatica or adrenal insufficiency, or asthma
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment (i.e. other investigational therapy, anti-neoplastic therapy, etc.) for their cancer
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
  * Nursing women - NOTE: breastfeeding should be discontinued if the mother is treated with nab-paclitaxel (Abraxane®)
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 28 days after stopping treatment
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Patients with a >= grade 2 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11-05; Primary Completion 2015-01-15 (Actual); Study Completion 2015-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fonseca, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy): Patients receive 100 mg nab-paclitaxel IV over 30 minutes on days 1, 8, and 15 (with 1 week rest). Treatment repeats every 28 days for up to 12 courses/cycles in the absence of disease progression or unacceptable toxicity. After 12 cycles, continued treatment is at the discretion of the investigator until evidence of disease progression. Paclitaxel Albumin-Stabilized Nanoparticle Formulation: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 70.0 [46.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have a Confirmed Partial Response or Better
Description: A confirmed partial response or better will be considered synonymous with "success" and is defined to be a stringent complete response (sCR = complete response (CR) + Normal serum FLC ratio + Absence of clonal cells in bone marrow), CR (= Negative immunofixation of the serum and urine + <5%plasma cells in bone marrow + Disappearance of any soft tissue plasmacytomas + normalization of FLC ratio), very good partial response (VGPR = partial response (PR) + Serum and urine M-component detectable by immunofixation but not on electrophoresis ), or PR (≥ 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24 h) noted as the objective status on two consecutive evaluations. The percentage of successes (confirmed PR or better) will be estimated by the number of successes divided by the total number of evaluable patients times 100. Confirmed PR or better will be evaluated using all cycles of treatment.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
percentage of patients | 7.7 [0.19 to 36]

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
months | 3.7 [1.7 to NA] — The upper limit of the 95% confidence interval was not reached.

3. Secondary Outcome: Progression Free Survival at 3 Months
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier and the 3 month progression-free rate (percentage) will be provided. Progression is defined as:
  Any one or more of the following: Increase of 25% from lowest value in:
  * Serum M-component (absolute increase must be ≥ 0.5 g/dl
  * Serum M-component increase ≥ 1 g/dl, if lowest M component was ≥ 5 g/dl
  * Urine M-component (absolute increase must be ≥ 200 mg/24 h)
  * If at on study, the only measurable non-bone marrow parameter was free light chain (FLC), the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dl)
  * Bone marrow plasma cell percentage (absolute % must be ≥10%) Or any one or more of the following felt related to the underlying clonal plasma cell proliferative disorder
  * Development of new soft tissue plasmacytomas or bone lesions
  * Hypercalcemia (≥11.5 mg/dl)
  * Decrease in hemoglobin of ≥2 g/dl
  * Serum creatinine level ≥2 mg/dl
Time Frame: Time from registration to the earliest date of documentation of disease progression, assessed up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
percentage of patients | 25.4

4. Secondary Outcome: Duration of Response of All Evaluable Patients Who Have Achieved a Partial Response or Better
Description: Duration of response is defined for all evaluable patients who have achieved a partial response or better (stringent complete response (sCR = complete response (CR) + Normal serum FLC ratio + Absence of clonal cells in bone marrow), CR (= Negative immunofixation of the serum and urine + <5%plasma cells in bone marrow + Disappearance of any soft tissue plasmacytomas + normalization of FLC ratio), very good partial response (VGPR = partial response (PR) + Serum and urine M-component detectable by immunofixation but not on electrophoresis ), or PR (≥ 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24 h) ) as the date at which the patients earliest best objective status is first noted to be at least a partial response or better to the earliest date of progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: Date at which the patient's earliest best objective status is first noted to be at least a partial response or better to the earliest date progression is documented, assessed up to 3 years
Population: All evaluable patients who have achieved a (unconfirmed or confirmed) partial response or better at the earliest best objective status are included in this analysis
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 2
months | 2.43 [NA to NA] — The lower and upper limits of the full range are not reported to avoid identification of individuals.

5. Secondary Outcome: Incidence of Toxicity as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The percentage of patients with a maximum grade 3 or higher adverse event at least possibly related to the study treatment are reported below.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
percentage of patients
  White blood cell decreased | 30.8
  Neutrophil count decreased | 38.5
  Platelet count decreased | 38.5
  Fatigue | 23.1
  Anemia | 15.4
  Anorexia | 7.7
  Edema limbs | 7.7
  Hyponatremia | 15.4
  Epistaxis | 7.7
  Febrile neutropenia | 7.7
  Infections and infestations | 7.7
  Lung infection | 7.7

6. Secondary Outcome: Overall Response Rate
Description: Overall response rate (percentage) is defined as the percentage of patients with a partial response (PR) or better. A PR or better will be considered synonymous with "success" and is defined to be a stringent complete response (sCR = complete response (CR) + Normal serum FLC ratio + Absence of clonal cells in bone marrow), CR (= Negative immunofixation of the serum and urine + <5%plasma cells in bone marrow + Disappearance of any soft tissue plasmacytomas + normalization of FLC ratio), very good partial response (VGPR = PR + Serum and urine M-component detectable by immunofixation but not on electrophoresis ), or PR (≥ 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24 h) noted as the objective status. The percentage of successes (PR or better) will be estimated by the number of successes divided by the total number of evaluable patients times 100. PR or better will be evaluated using all cycles of treatment.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 13
percentage of patients | 15 [1.9 to 45.5]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored within 14 days prior to registration, prior to subsequent treatment (visits at the end of each cycle), and at end of treatment, assessed up to 3 years.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Treatment (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 11/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=13)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophageal necrosis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=13)
Anemia (Blood and lymphatic system disorders) | 7 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (14)
Nausea (Gastrointestinal disorders) | 7 (10)
Edema limbs (General disorders) | 1 (3)
Fatigue (General disorders) | 13 (28)
Fever (General disorders) | 5 (7)
Malaise (General disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (6)
Neutrophil count decreased (Investigations) | 11 (18)
Platelet count decreased (Investigations) | 7 (11)
White blood cell decreased (Investigations) | 13 (23)
Anorexia (Metabolism and nutrition disorders) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (26)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (11)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes